CLINICAL TRIAL: NCT06274996
Title: A Retrospective Analysis of the Efficacy and Safety of Upadacitinib in the Treatment of Inflammatory Bowel Disease
Brief Title: Efficacy and Safety Analysis of Upadacitinib in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiayin Yao, Associate Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2024ZSLYEC-063
Record Dates: First submitted 2024-02-03; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib, a selective Janus kinase (JAK) inhibitor taken orally, is being assessed for its unique capacity to attenuate inflammatory pathways in IBD at a cellular level by selectively inhibiting JAK1, a pathway integral to inflammatory cytokine production. This study focuses on its use as monotherapy for Chinese patients unresponsive to conventional IBD treatments, such as aminosalicylates and corticosteroids. By centering on a demographic typically underrepresented in research, the study aims to provide new insights into dosing, treatment frequency, and duration, thus enhancing the understanding of Upadacitinib's safety and efficacy. The retrospective analysis of patient data is anticipated to inform more personalized treatment approaches, potentially improving IBD management and patient quality of life.

SUMMARY:
This study focuses on evaluating Upadacitinib, a new oral medication that inhibits specific enzymes involved in inflammation, for treating inflammatory bowel disease (IBD), which includes conditions such as Crohn's Disease and Ulcerative Colitis. The goal is to determine how effective and safe this drug is for patients in China, where data is currently lacking.IBD significantly affects individuals' quality of life and imposes a high burden on society and healthcare systems. Current treatments don't work for everyone, and some patients may need surgery. Upadacitinib has shown promise in other countries for treating IBD and related conditions and has been approved by the US FDA for such use.

Our study is retrospective and multicenter, meaning it will look back at patient records from multiple hospitals to analyze the outcomes of those who have received Upadacitinib. Investigators aim to enroll patients treated between January 2020 and December 2023, focusing on adults who have taken Upadacitinib for at least 8 weeks.For patients, families, and healthcare providers, this research could mean a potential new treatment option for IBD. Understanding Upadacitinib's efficacy and safety could lead to better management of the disease, possibly reducing the need for surgery and improving the quality of life for those affected by IBD. The ultimate goal is to provide more personalized and effective treatment strategies for IBD patients in China.

DETAILED DESCRIPTION:
This retrospective, multicenter study is designed to evaluate the efficacy and safety of Upadacitinib, an oral selective enzyme inhibitor, in the treatment of inflammatory bowel disease (IBD) within the Chinese patient population. IBD, encompassing conditions such as Crohn's Disease and Ulcerative Colitis, poses a significant impact on the quality of life for individuals and presents a considerable challenge to healthcare systems due to the societal burdens it incurs. While current therapeutic interventions offer relief, they fail to suffice for all patients, with some requiring surgical intervention. Despite the approval of Upadacitinib by the US FDA and its promising application in other nations for IBD management, there is a scarcity of data on its effectiveness and safety among Chinese patients.Our research aims to fill this knowledge gap by retrospectively analyzing patient records from multiple hospitals across China. The study targets the adult patient demographic that has undergone Upadacitinib treatment for a minimum duration of eight weeks between January 2020 and December 2023. By assessing the outcomes of these patients, our objective is to ascertain the potential of Upadacitinib as a viable treatment alternative, which may revolutionize the current IBD treatment paradigm in China.

The implications of this study are significant for patients, their families, and healthcare providers, as it could herald a new therapeutic avenue for IBD management. A clearer understanding of Upadacitinib's role in disease control could enhance patient care by decreasing the necessity for surgical procedures and ameliorating life quality for IBD sufferers. The overarching ambition of this research is to pave the way for more individualized and efficacious treatment methodologies for the IBD patient populace in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized in our institution or its branches between January 2020 and September 2023.

Patients with a confirmed diagnosis of Crohn's Disease (CD) or Ulcerative Colitis (UC).

Patients aged 18 years or older. Patients who have received at least 8 weeks of Upadacitinib treatment prior to December 2023.

Exclusion Criteria:

* Patients with an unclear diagnosis. Patients under the age of 18. Patients who have been treated with Upadacitinib for less than 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients aged 18 and older who were hospitalized for Crohn's Disease (CD) or Ulcerative Colitis (UC) between January 2020 and September 2023 at our institution or its branches, and who have been treated with Upadacitinib for at least 8 weeks prior to December 2023. The focus is on adults with a confirmed diagnosis to assess the treatment's efficacy in inducing clinical remission and altering disease progression. Exclusion criteria include unclear diagnosis, patients under 18, and Upadacitinib treatment for less than 8 weeks, ensuring a uniform group for valid results.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Steroid-Free Clinical Remission | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8weeks and up to 24 weeks
  Clinical remission in CD is defined as a CDAI score of less than 150, achieved without the use of corticosteroids.Clinical remission in UC is defined as a modified Mayo score of 2 or less, with no individual subscore greater than 1, achieved without the use of corticosteroids.

SECONDARY OUTCOMES:
Clinical Response | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8 weeks and up to 24 weeks
  CD:A decrease in CDAI score by 70 points or more from baseline is considered a clinical response. UC: A decrease in the Modified Mayo Score by at least 30% and an absolute reduction of at least 3 points from baseline signifies a clinical response.
Endoscopic Remission | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8 weeks and up to 24 weeks
  CD:An SES-CD score of 2 or less indicates endoscopic remission. UC: An MES of 1 or less is defined as endoscopic remission.
Mucosal Healing | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8 weeks and up to 24 weeks
  CD:An SES-CD score of 0 is indicative of mucosal healing. UC:An MES of 0 represents mucosal healing.
Radiological remission | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8 weeks and up to 24 weeks
  Defined as the complete disappearance or minimization of intestinal inflammation on imaging studies, signifying no visible lesions, normalized wall thickness, absence of strictures or obstructions, and no new areas of disease. Radiographic remission is an important indicator of deep remission in disease treatment goals.
Radiological response | CD:Assessed at 12 weeks and up to 24 weeks; UC：Assessed at 8 weeks and up to 24 weeks
  Typically defined as a significant reduction in the size of affected areas, decreased wall thickness, and decreased markers of inflammation observed through imaging methods such as MRI or CT scans. A radiographic response indicates a reduction in disease activity but may not represent complete disease remission.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No